CLINICAL TRIAL: NCT06317259
Title: Impacts of Rhythmic and Hypoxic Breathwork on EEG, Mood, Sleep, and Physiology
Brief Title: Effects of Hypoxic Breathwork
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Julie Onton, Project Scientist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 809163
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hypoxic Breathwork With Music and Affirmative Messaging; Hypoxic Breathwork Only; Music and Affirmative Messaging
Keywords: Breathwork; Intermittent hypoxia; EEG; Mitochondria; Relaxing

STUDY DESIGN:
Intervention Model Description: We have 3 groups running in parallel (one of each group running in the same week). Group 1 will do breathwork that includes music and positive messaging, group 2 will do breathwork alone with only guided breathing instructions, and group 3 will listen to the music and positive messaging but no breathwork which we call the "meditation" group.
Who Masked: Participant
Masking Description: Subjects will be unaware of the other conditions and will thus not know if they are in a 'control' group or not. All experimenters will know subject group assignments. Subjects will be told of all groups at the end.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathwork, music, messaging (Experimental): Subjects will perform a 40 min initial breathwork/music/messaging session with a full EEG cap followed by 7 or 14 days of once daily practice of a 20 min breathwork/music/messaging session. At the end of 7 or 14 days, they will again perform the 40 min breathwork/music/messaging session with a full EEG cap.
  Interventions: Behavioral: Hypoxic breathwork plus music and messaging
- Breathwork only (Active Comparator): Subjects will perform a 40 min initial breathwork only session with a full EEG cap followed by 7 or 14 days of once daily practice of a 20 min breathwork only session. At the end of 7 or 14 days, they will again perform the 40 min breathwork only session with a full EEG cap.
  Interventions: Behavioral: Hypoxic breathwork only
- Music and messaging (Active Comparator): Subjects will perform a 40 min initial music/messaging session with a full EEG cap followed by 7 or 14 days of once daily practice of a 20 min music/messaging session. At the end of 7 or 14 days, they will again perform the 40 min music/messaging session with a full EEG cap.
  Interventions: Behavioral: Music and messaging meditation

INTERVENTIONS:
Behavioral: Hypoxic breathwork plus music and messaging — Hypoxic breathwork consists of about 5 min of rhythmic breathing in a 4-in/4-out pattern followed by a breath hold on the exhale for about 1-2 min. This is repeated 1-2 times with increasing breath rate up to 2-in/2-out. The audio track also includes dynamic music that accompanies the different stages as well as positive messaging encouraging self-determination.
  Arms: Breathwork, music, messaging
Behavioral: Hypoxic breathwork only — Hypoxic breathwork consists of about 5 min of rhythmic breathing in a 4-in/4-out pattern followed by a breath hold on the exhale for about 1-2 min. This is repeated 1-2 times with increasing breath rate up to 2-in/2-out. Other than breathing instructions and pacing, the audio track is silent.
  Arms: Breathwork only
Behavioral: Music and messaging meditation — Music and messaging meditation consists of dynamic music that is engaging and aids focus, as well as positive messaging encouraging self-determination.
  Arms: Music and messaging

SUMMARY:
This project will study changes that occur during a short period of intensive daily slow-paced breathing and breath hold practice (i.e., "breathwork"). On the first and last days of the week-long practice, investigators will conduct high-density EEG recordings during breathwork to evaluate spectral power, coherence, and causality dynamics of the brain when it is naïve to breathwork and after adaptation to a breathwork practice. Breath, blood, urine, saliva, stool samples, biometric data, and sleep EEG will be collected before the start of daily breathwork practice and again after 1 week of breathwork practice to examine the effect of breathwork on full body biochemistry, molecular biology, and sleep. Investigators will also use questionnaires to assess the impact of breathwork on stress and sleep quality.

DETAILED DESCRIPTION:
Breathwork. Breathwork simply means consciously manipulating the breath to achieve a desired result. There are many kinds of breathwork for different goals. An entire segment of yoga, called pranayama, harnesses the power of breath manipulation for various health benefits. The current study does not use a specific technique from ancient traditions but combines two basic techniques grounded in Western literature: slow-paced breathing and hypoxic breath-hold training.

Breathwork: slow-paced breathing. The study of slow-paced breathing (SPB) emerged from the observation that heart rate follows the breath: heart rate increases during inhale and decreases during exhale. Multiple physiological processes come into alignment when breathing is maintained at a constant rate of about 0.1 Hz (6 breaths per minute). Since slower breathing necessitates larger tidal volume, SPB causes rhythmic changes in blood pressure, which triggers the baroreflex response. The baroreflex involves communication from the body to the brain stem and higher brain centers via vagal nerve afferents. The brain projects back through the vagus nerve to the heart, releasing acetylcholine, to cause temporary heart slowing. Because typical breath (in our culture anyway) is usually much faster and less regular, this resonance is not achieved in normal daily living, leading to reduced parasympathetic function. Practicing SPB can help to restore health by recovery of proper autonomic balance. For example, blood pressure is acutely reduced during SPB, along with increased baroreflex sensitivity. Systolic blood pressure was reduced in hypertensive patients after 8 and 12 weeks of SPB practice. It can also reduce blood pressure and increase oxygen absorption in sea level dwellers exposed to high altitudes.

In addition to brain stem targets of vagal afferents, dorsal pons, periaqueductal grey matter, cerebellum, hypothalamus, thalamus, and lateral and anterior insular cortices also show activity on functional magnetic resonance imaging (fMRI) during SPB (Critchley et al., 2015). A regular practice of SPB for 8 weeks has also been shown to increase functional connectivity between the ventromedial prefrontal cortex and the insula, amygdala, middle cingulate, and lateral prefrontal cortex compared to controls (Schumann et al., 2021).

Breathwork: breath hold. Various research avenues have shown the surprising benefits of intermittent low oxygen. Throughout the ages, different cultures have had some level of awareness about breathing less or moving to altitude for health reasons. Specific studies began to be performed when humans began high altitude activities like hot air ballooning and mountaineering and from there many discoveries have been made about the benefits of low oxygen. For example, high altitude living for athletes confers advantages for training and competition at sea level, and yogi masters have taught pranayama (breathing techniques) that limit oxygen exposure for various benefits like stress reduction or clearing the mind. But these are only the most obvious sequelae of lowered oxygen. More surprising is that hypoxic preconditioning protects against subsequent ischemic challenge that would normally result in neuronal death. Reduced oxygen has also been shown to boost growth factors, increase neurogenesis, improve blood flow to the brain and increase antioxidant activity. The mechanism of such benefits is thought to mostly involve hypoxia-inducible factors (HIFs), which lead to downstream effectors such as heme-oxygenase-1, heat-shock proteins, growth factors, erythropoietin and more. Thus, as counter-intuitive as it might seem, limiting oxygen, either by reduced oxygen gas mixtures, altitude, or breath-holding, is an effective way to stimulate the body's natural abilities to increase health-promoting factors.

EEG brain imaging of breathwork. In this study, we will use a 128-channel EEG cap to record whole-head EEG that will allow for decomposition into cortical source activity using independent component analysis (ICA). This technique has the advantage of separating activities emanating from different areas of the brain (instead of scalp locations) and then observing their transient interactions during specific tasks. In this study, we will examine source activity during guided rhythmic breathing and breath-hold sequences to observe the frequency power and coherences that characterize these states. The effect of hypoxia on the EEG has not been extensively studied, and preliminary reports are varied, partly because of varied techniques for inducing hypoxia. For example, hypobaric hypoxia has been shown to increase in alpha (~8-12 Hz) and theta (~4-7 Hz) frequencies in one study, but decrease alpha in two other studies, though these both did find a consistent increase in theta power. Normobaric breath holding has also been shown to decrease alpha activity. Furthermore hypercapnia, or increased carbon dioxide (CO2) (which also occurs during breath hold), has also been noted to decrease alpha, as well as beta (~13-30 Hz) and low gamma (~30-50 Hz) using magnetoencephalography.

SPB also has a small literature showing spectral changes during and after controlled breathing. One study of a specific pranayama technique showed a theta increase during SPB which drops during subsequent meditation, while alpha power decreased during SPB and decreased further during meditation. Using a different experimental design, another study showed progressive increases in total power and all spectral bands (theta, alpha, beta) when subjects performed rapid breathing, normal breathing, and SPB. However, another study found decreased low beta power during SPB as compared to rapid breathing. SPB has also been shown to synchronize slow cortical potentials and heart rate variability (HRV), leading to a subjectively relaxing state for subjects.

While these reports show clear evidence for EEG changes during voluntary breath manipulation, their results are both inconsistent and using only the most basic analysis techniques. In the current study, we intend to extend these findings by decomposing the high-density EEG data into independent components using ICA and examine the coherence and causality of the EEG activity to show the level of brain connectedness and directions of information flow during these states of altered consciousness.

Physiology, Biochemistry, and Molecular Biology. No studies have been undertaken to integrate the physiological, biochemical, and molecular biological responses of breathwork in humans. Studies have assessed transcriptome changes during Yoga that show main effects on immune modulation, but these are complicated by processes that include breathwork in addition to other manipulations. Ours will be the first study to integrate multiple physiological and biological multi-omic endpoints to study the impact of breath training.

ELIGIBILITY:
Inclusion Criteria:

* Persons, aged 18-45
* Availability for the duration of the study
* In good general health as revealed by self-report
* Stated willingness and capability to adhere to the breathwork regimen
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration
* Provision of signed and dated informed consent form

Exclusion Criteria:

1. Current or past regular breathwork practice
2. Current use of psychoactive medications (e.g., anti-depressants or anxiolytics)
3. Pregnancy
4. Bedtime past 11:30pm or regularly getting less than 6 hours of sleep per night.
5. Feverish illness within 10 days
6. Regular smoker or tobacco user ( > 1 cigarette, gum or pouch per month)
7. Presence of blood pressure above 140 systolic and/or 90 diastolic, seizure disorder, asthma, or serious cardiac fibrillation disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EEG power and/or connectivity differences between groups | Day 7 and Day 14 or 21 (beginning and end of daily practice week)
  EEG features will be extracted to show the brain responses to rhythmic breathing and hypoxic breath holds that will be compared with music and positive messaging meditation. These groups will also be compared with a breathwork only condition.
Group differences in sleep EEG power and/or stage changes from baseline to the intervention period | Days 7-14 or 21 (intervention) vs Days 1-7 (baseline)
  Sleep stages and power characteristics will be analyzed during the practice week as compared to the week prior during which they have no intervention. All three experimental groups will be compared.

SECONDARY OUTCOMES:
Group differences between physiological changes in proteomics, microbiome, and other factors from baseline following intervention | Days 1 and 14 or 21 (before and after intervention)
  Physiological factors from blood, urine, saliva, stool and breath will be compared from before to after the 7-day intervention.
Group differences in mood and stress from before to after the intervention | Days 1 and 14 or 21 (before and after intervention)
  Subjects will report their mood, sleep and stress levels before and after the intervention. All experimental groups will be compared.
  Insomnia Severity Index (0-no sleep problems to 28-very severe sleep problems) ; Perceived Stress Questionnaire (0-no stress to 40-high stress) ; Mystical Experiences-30 (0-no mystical feelings to 150-extreme mystical feelings) ; PROMIS-29 (5 subscales: Fatigue/SleepDisturbance/PainInterference range from 20-80 with 80 being the more severe; Ability to participate in social roles and activities ranges from 80-20 with 20 being more severe disruption; Pain Intensity ranges from 0-10 with 10 being the worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data with anyone outside of the current study staff.